CLINICAL TRIAL: NCT06966856
Title: Sublingual Versus Oral Vitamin B12 for Acute Hypovitaminosis B12 Secondary to Proton Pump Inhibitors: A Prospective Randomized Study
Brief Title: This Randomized, Clinical Trial Evaluates the Efficacy of Oral Versus Sublingual Vitamin B12 Supplementation in Correcting Early-onset Vitamin B12 Deficiency in Adult Patients Using Proton Pump Inhibitors (PPIs). The Primary Outcome is the Change in Serum Vitamin B12 Levels Over a 6-week
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reem Alaa Abdel Samie, teacher assistant in Delta University for science and technology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORSUB12
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Hypovitaminosis b 12
MeSH Terms: interventions — Vitamin B 12; Tablets; Administration, Sublingual; Omeprazole; Esomeprazole; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Vitamin B12 Group (Experimental): Participants in this arm will receive 1000 mcg oral cyanocobalamin daily for 6 weeks. The supplement will be administered as a swallowed tablet. Patients will continue their regular PPI therapy during the study period.
  Interventions: Drug: Cyanocobalamin 1000 Mcg Oral Tablet
- Sublingual Vitamin B12 Group (Experimental): Participants in this arm will receive 1000 mcg sublingual cyanocobalamin daily for 6 weeks. The supplement will be administered as a sublingual tablet placed under the tongue. Patients will continue their regular PPI therapy during the study period.
  Interventions: Drug: Cyanocobalamin 1000 Mcg Sublingual Tablet
- Control Group (PPI Only) (Active Comparator): Participants in this arm will continue their regular PPI therapy without receiving vitamin B12 supplementation. This arm serves as a control to evaluate natural changes in B12 levels without supplementation.
  Interventions: Other: Proton Pump Inhibitor therapy only

INTERVENTIONS:
Drug: Cyanocobalamin 1000 Mcg Oral Tablet — Oral cyanocobalamin supplement administered as a 1000 mcg tablet taken once daily for 6 weeks. Used in patients with early-onset B12 deficiency during PPI therapy.
  Other Names: Vitamin B12 tablet (oral)
  Arms: Oral Vitamin B12 Group
Drug: Cyanocobalamin 1000 Mcg Sublingual Tablet — Sublingual cyanocobalamin supplement administered as a 1000 mcg tablet placed under the tongue once daily for 6 weeks. Used in patients with early-onset B12 deficiency during PPI therapy.
  Other Names: Sublingual vitamin B12, B12 lozenge, Methylcobalamin sublingual
  Arms: Sublingual Vitamin B12 Group
Other: Proton Pump Inhibitor therapy only — This group will continue their standard PPI therapy without receiving any vitamin B12 supplementation, serving as a control group for the comparison of B12 correction efficacy.
  Other Names: PPI, omeprazole, esomeprazole, pantoprazole
  Arms: Control Group (PPI Only)

SUMMARY:
This randomized, clinical trial evaluates the efficacy of oral versus sublingual vitamin B12 supplementation in correcting early-onset vitamin B12 deficiency in adult patients using proton pump inhibitors (PPIs). The primary outcome is the change in serum vitamin B12 levels over a 6-week treatment period. Secondary outcomes include changes in homocysteine levels, hemoglobin levels, and patient-reported satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70.
* PPI use for 1-6 months (new users).
* Serum B12 between 150-300 pg/mL.
* No known prior B12 supplementation.

Exclusion Criteria:

* History of long-term GI disease (e.g., Crohn's, celiac).
* Previous gastrectomy/bariatric surgery.
* Baseline anemia with hemoglobin <9 g/dL.
* Severe renal or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Vitamin B12 Concentration | Baseline and Week 6
  Measurement of serum vitamin B12 levels before and after 6 weeks of intervention to assess the efficacy of oral versus sublingual supplementation.

SECONDARY OUTCOMES:
Change in Plasma Homocysteine Level | Baseline and Week 6
  Plasma homocysteine levels will be measured at baseline and at 6 weeks to assess the functional improvement in vitamin B12 status.
Change in Hemoglobin Level | Baseline and Week 6
  To assess improvement in anemia, hemoglobin concentration will be measured at baseline and at 6 weeks.
Patient-Reported Satisfaction with Route of Supplementation | Week 6
  At the end of the study, patients will be surveyed about their satisfaction and ease of use with the assigned supplementation route (oral or sublingual).